CLINICAL TRIAL: NCT06464380
Title: Anti Cancer Potential of Saffron in Hepatocellular Carcinoma
Brief Title: Anti-cancer Potentiality of Saffron Against Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Amr Amin College of Medicine, University of Sharjah, Sharjah 27272, UAE. (Unknown); Ahmed Cordie Endemic Medicine department, Cairo University Hospitals. (Unknown); Nouran Mohamed Endemic Medicine department, Cairo University Hospitals. (Unknown); Gamal Esmat Faculty of Biotechnology, Misr University for Science and Technology, Giza, Egypt. (Unknown)
Responsible Party: Principal Investigator, Amal A. Elkholy, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1167/05/2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Saffron
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant
Masking Description: Single blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- safranal Group (Active Comparator): include 20 HCC patients will receive 50 mg safranal regimen in dose of once per day for six months.
  Interventions: Dietary Supplement: Saffranal
- Control Group (Placebo Comparator): include 20 HCC patients will receive placebo in the form of once per day for six months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saffranal — HCC patients will receive 50 mg safranal regimen in dose of once per day for six months.
  Arms: safranal Group
Dietary Supplement: Placebo — HCC patients will receive Placebo in dose of once per day for six months.
  Arms: Control Group

SUMMARY:
Saffron has recently gained considerable interest for its capacity to interfere with cancer at initiation and promotion stages as well as for cancer treatment. Although saffron and its constituents have been shown to have antitumorigenic and proapoptotic activities in different cancer cell lines.

The aim of the current investigation is to identify the anti-cancer potentiality of saffron on hepatocellular carcinoma patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer and the third leading cause of cancer mortality in the world. Chronic infection with hepatitis B and C is the major risk factors for HCC worldwide. Other factors that contribute to the formation of HCC include exposure to environmental carcinogens, iron overload, fatty liver disease, and alcohol abuse.

there has been a sustained rise in its incidence in both developing and developed countries. Despite the growing therapeutic options for patients with cancer, their efficacy is time-limited and non-curative. Hence to overcome these drawbacks, an incessant screening for superior and safer drugs has been ongoing for numerous decades, resulting in the detection of anti-cancer properties of several phytochemicals. Chemoprevention using readily available natural substances from vegetables, fruits, herbs and spices is one of the significantly important approaches for cancer prevention in the present era. Among the spices, saffron has generated interest because pharmacological experiments have established numerous beneficial properties including radical scavenging, anti-mutagenic and immuno-modulating effects.

Saffron is a naturally derived plant product from the dried stigma of the Crocus sativus flower (family Iridaceae) that may have biologically useful properties. In fact, saffron extract and its biologically active compounds, including crocin, crocetin, carotene, and safranal, have been shown both in vitro and in vivo to possess antioxidant, anticancer, anti-inflammatory, and memory-improving properties. Saffron is also used in folk medicine as an antispasmodic, antidepressant, and aphrodisiac. Furthermore, it is one of the most commonly used species around the world for flavouring and colouring foods.

Saffron has recently gained considerable interest for its capacity to interfere with cancer at initiation and promotion stages as well as for cancer treatment. Although saffron and its constituents have been shown to have antitumorigenic and proapoptotic activities in different cancer cell lines.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients above 18 years
* Patients with end-stage HCC not candidate for curative, loco regional treatment and /or systemic chemotherapy
* Patients with available baseline laboratory parameters and contrast- enhancing images after given written consent for research participation.

Exclusion Criteria:

* Patients who are candidate for curative and/or loco-regional or combination treatment for HCC
* Patients with concomitant malignancies other than HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | three months
  overall survival in patients presented with end-stage hepatocellular carcinoma.

SECONDARY OUTCOMES:
treatment response | three months
  response to treatment through impact on the underlying liver status

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Amal A. Elkholy, Al ‘Abbāsīyah, Al Abbasiya
  - Dermatology Clinic of National Hepatology and Tropical Medicine Research Institute, Cairo

REFERENCES:
- [Background] Abdullaev FI, Espinosa-Aguirre JJ. Biomedical properties of saffron and its potential use in cancer therapy and chemoprevention trials. Cancer Detect Prev. 2004;28(6):426-32. doi: 10.1016/j.cdp.2004.09.002. PMID 15582266
- [Background] Abdullaev FI. Cancer chemopreventive and tumoricidal properties of saffron (Crocus sativus L.). Exp Biol Med (Maywood). 2002 Jan;227(1):20-5. doi: 10.1177/153537020222700104. PMID 11788779
- [Background] Bhandari PR. Crocus sativus L. (saffron) for cancer chemoprevention: A mini review. J Tradit Complement Med. 2015 Jan 28;5(2):81-7. doi: 10.1016/j.jtcme.2014.10.009. eCollection 2015 Apr. PMID 26151016
- [Background] Das I, Das S, Saha T. Saffron suppresses oxidative stress in DMBA-induced skin carcinoma: A histopathological study. Acta Histochem. 2010 Jul;112(4):317-27. doi: 10.1016/j.acthis.2009.02.003. Epub 2009 Mar 27. PMID 19328523